CLINICAL TRIAL: NCT05416099
Title: Comparing Conventional Grid Laser Photocoagulation and Subthreshold Micropulse Laser in Diabetic Macular Edema Using OCT Angiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anita Li, Dr, Chinese University of Hong Kong
Other Study IDs: gridvsmicropulseDMEOCTA
Record Dates: First submitted 2022-06-03; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grid laser: grid laser is one of the more conventional treatments for diabetic macular edema
  Interventions: Procedure: laser
- micropulse laser: micropulse laser is one of the more recent treatments for diabetic macular edema
  Interventions: Procedure: laser

INTERVENTIONS:
Procedure: laser — grid vs micropulse laser

SUMMARY:
The prevalence of diabetes mellitus has increased significantly in Hong Kong for the past decade [1]. Diabetic macular edema is one of the most common causes of vision loss in patients suffering from diabetes mellitus [3]. Before the introduction of anti-vascular endothelial growth factor agents, laser photocoagulation has been the mainstay treatment for patients with diabetic macular edema. There are two types of laser treatment modalities, namely focal laser, which can be applied either in a grid pattern over a region of macular edema or to selected microaneurysms, and subthreshold micropulse laser. Only one meta-analysis published in 2016 [16] had previously demonstrated superiority of micropulse laser over focal laser, while other studies showed no clinically significant differences between the two lasers. Nevertheless, micropulse laser had been proven to cause no structural changes to the retina and choroid, as opposed to focal laser.

Optical coherence tomography angiography (OCT-A) is a new, non-invasive imaging technique that allows a clear, depth-resolved visualization of the retinal and choroidal microvasculature in the macular region [22]. A recent case series study [17] has demonstrated early changes of retinal vasculature on OCT-A images after micropulse laser for diabetic macular edema. Another cross-sectional study [18] showed choriocapillaries alterations in some of the patients after receiving focal laser. We would like to compare the changes of different OCT-A parameters for patients receiving either type of laser, and hence evaluating their efficacy.

We propose to take OCT-A images for patients before laser, 1-, 3- and 6-months post-laser based on the results of a recent case series [17]. We will analyse the OCT-A images with MATLAB software and compare the changes in different parameters between both lasers.

DETAILED DESCRIPTION:
Laser photocoagulation was previously a mainstay treatment for DME before the introduction of anti-vascular endothelial growth factor (anti-VEGF) agents injection. Vascular endothelial growth factor (VEGF) is an important mediator of blood-retinal barrier breakdown, which leads to fluid leakage and the development of macular edema [5]. Observing that intraocular VEGF levels are increased in DME, using VEGF inhibitors (anti-VEGF) was found to be beneficial in reversing vision loss from macular edema [6]. In recent years, many large-scale studies [7], [8], [9], [10] had proven that anti-VEGF injections resulted in superior improvements in visual acuity and central subfield thickness than laser photocoagulation in treating DME. This has led to the decline of conventional focal laser as a first-line therapy.

However, in our clinical setting, laser photocoagulation may still be preferred in selected clinical scenarios in treating DME. In Hong Kong, anti-VEGF agents were self-financed items for patients in the public sector of our healthcare system. These medications could be a huge financial burden to patients with low financial support, and therefore they might prefer laser therapy instead.

Furthermore, anti-VEGF intravitreal injections have been reported to have detectable levels in systemic circulation, which can lead to systemic complications. A retrospective study [11] of 1173 patients showed that bevacizumab has a risk of leading to systemic events including acute blood pressure elevation (0.59%), cerebrovascular accidents (0.5%), myocardial infarctions (0.4%), and iliac artery aneurysms (0.17%). Hence, patients with recent history of cardiovascular accidents or significant cardiovascular comorbidities and patients who could not tolerate intravitreal injections might also find laser therapy a better option in treating DME.

Therefore, it is still useful to compare the effectiveness of conventional focal/grid laser versus subthreshold micropulse in treating DME in our clinical context. Previous studies [12], [13], [14] had mainly demonstrated non-inferiority of subthreshold micropulse laser in terms of best-corrected visual acuity (BCVA), contrast sensitivity and central retinal thickness. Nonetheless, majority of the studies demonstrated that laser scars were much more frequently identified in conventional laser than micropulse laser-treated eyes.

Optical coherence tomography angiography (OCT-A) is a new, non-invasive imaging technique to visualize the retinal vasculature and choroidal vascular layers in the macular area. It employs motion contrast imaging to high-resolution volumetric blood flow information, generating angiographic images in seconds. The principle of OCT-A involves the comparison of decorrelation signal between sequential Optical Coherence Tomography (OCT) B-scans taken at precisely the same cross-section, therefore constructing a map of blood flow. Given that only erythrocyte movements in the blood vessels are represented and axial bulk motions are eliminated, determining a vascular decorrelation signal enables visualization of 3-dimensional retinal and choroidal vascular network without the administration of intravenous dye and thus reducing the risk of potential adverse events [17], [22].

The authors believe that OCT-A can be used as a new assessment tool in comparing the efficacy of conventional focal laser versus subthreshold micropulse laser in the treatment of DME. We hypothesize that subthreshold micropulse laser is superior to focal laser in treating patients with DME in terms of OCT-A parameters. We expect the reduction in the studied OCT-A parameters (i.e. FAZ area, area of cysts, number of microaneurysms, etc.) in patients receiving subthreshold micropulse laser will be greater than focal laser by 30%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with best-corrected visual acuity better than 20/200 (checked with refraction test)
* Patients with clinically significant diabetic macular edema (DME) who have not received any treatment within 6 months
* Patients with central retinal thickness equal / above to around 400 um
* Patients who are able to have regular visits after laser treatment for at least 6 months

Exclusion Criteria:

* Children under the age of 18
* Patients with proliferative diabetic retinopathy
* Patients with co-existing retinal or macular disease, including epiretinal membrane and vitreomacular traction
* Patients with previous history of laser photocoagulation, anti-VEGF injection, intravitreal steroid injection, vitreoretinal or cataract surgery within a period of 6 months
* Patients with history of uveitis
* Patients who are unfit or for capturing of OCT-A images
* Patients with significant media opacity that may interfere with fundal examination and the acquisition of high quality OCT-A images
* Patients who are unable to give informed consent to enter the study

uncooperative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic macular edema and central retinal thickness >400micrometers who have not received any treatments within 6 months
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity | 1 month, 3 month and 6 months

SECONDARY OUTCOMES:
Change in OCTA parameters | 1 month, 3 month and 6 months
  Change in OCT measurement of FAZ area

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel HK Li, M.B. Ch.B, Principal Investigator — CUHK
Locations (1):
- chinese university of Hong kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quan J, Li TK, Pang H, Choi CH, Siu SC, Tang SY, Wat NMS, Woo J, Johnston JM, Leung GM. Diabetes incidence and prevalence in Hong Kong, China during 2006-2014. Diabet Med. 2017 Jul;34(7):902-908. doi: 10.1111/dme.13284. Epub 2016 Nov 29. PMID 27859570
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Bandello F, Battaglia Parodi M, Lanzetta P, Loewenstein A, Massin P, Menchini F, Veritti D. Diabetic Macular Edema. Dev Ophthalmol. 2017;58:102-138. doi: 10.1159/000455277. Epub 2017 Mar 28. PMID 28351052
- [Background] Wan KH, Chen LJ, Young AL. Screening and Referral of Diabetic Retinopathy: A Comparative Review of the Practice Guidelines. Asia Pac J Ophthalmol (Phila). 2013 Sep-Oct;2(5):310-6. doi: 10.1097/APO.0b013e31829df4a3. PMID 26107035
- [Background] Qaum T, Xu Q, Joussen AM, Clemens MW, Qin W, Miyamoto K, Hassessian H, Wiegand SJ, Rudge J, Yancopoulos GD, Adamis AP. VEGF-initiated blood-retinal barrier breakdown in early diabetes. Invest Ophthalmol Vis Sci. 2001 Sep;42(10):2408-13. PMID 11527957
- [Background] Funatsu H, Yamashita H, Noma H, Mimura T, Yamashita T, Hori S. Increased levels of vascular endothelial growth factor and interleukin-6 in the aqueous humor of diabetics with macular edema. Am J Ophthalmol. 2002 Jan;133(1):70-7. doi: 10.1016/s0002-9394(01)01269-7. PMID 11755841
- [Background] Nguyen QD, Shah SM, Heier JS, Do DV, Lim J, Boyer D, Abraham P, Campochiaro PA; READ-2 Study Group. Primary End Point (Six Months) Results of the Ranibizumab for Edema of the mAcula in diabetes (READ-2) study. Ophthalmology. 2009 Nov;116(11):2175-81.e1. doi: 10.1016/j.ophtha.2009.04.023. Epub 2009 Aug 22. PMID 19700194
- [Background] Mitchell P, Bandello F, Schmidt-Erfurth U, Lang GE, Massin P, Schlingemann RO, Sutter F, Simader C, Burian G, Gerstner O, Weichselberger A; RESTORE study group. The RESTORE study: ranibizumab monotherapy or combined with laser versus laser monotherapy for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):615-25. doi: 10.1016/j.ophtha.2011.01.031. PMID 21459215
- [Background] Ishibashi T, Li X, Koh A, Lai TY, Lee FL, Lee WK, Ma Z, Ohji M, Tan N, Cha SB, Shamsazar J, Yau CL; REVEAL Study Group. The REVEAL Study: Ranibizumab Monotherapy or Combined with Laser versus Laser Monotherapy in Asian Patients with Diabetic Macular Edema. Ophthalmology. 2015 Jul;122(7):1402-15. doi: 10.1016/j.ophtha.2015.02.006. Epub 2015 May 14. PMID 25983216
- [Background] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934
- [Background] Wu L, Martinez-Castellanos MA, Quiroz-Mercado H, Arevalo JF, Berrocal MH, Farah ME, Maia M, Roca JA, Rodriguez FJ; Pan American Collaborative Retina Group (PACORES). Twelve-month safety of intravitreal injections of bevacizumab (Avastin): results of the Pan-American Collaborative Retina Study Group (PACORES). Graefes Arch Clin Exp Ophthalmol. 2008 Jan;246(1):81-7. doi: 10.1007/s00417-007-0660-z. Epub 2007 Aug 3. PMID 17674014
- [Background] Figueira J, Khan J, Nunes S, Sivaprasad S, Rosa A, de Abreu JF, Cunha-Vaz JG, Chong NV. Prospective randomised controlled trial comparing sub-threshold micropulse diode laser photocoagulation and conventional green laser for clinically significant diabetic macular oedema. Br J Ophthalmol. 2009 Oct;93(10):1341-4. doi: 10.1136/bjo.2008.146712. Epub 2008 Dec 3. PMID 19054831
- [Background] Vujosevic S, Bottega E, Casciano M, Pilotto E, Convento E, Midena E. Microperimetry and fundus autofluorescence in diabetic macular edema: subthreshold micropulse diode laser versus modified early treatment diabetic retinopathy study laser photocoagulation. Retina. 2010 Jun;30(6):908-16. doi: 10.1097/IAE.0b013e3181c96986. PMID 20168272
- [Background] Lavinsky D, Cardillo JA, Melo LA Jr, Dare A, Farah ME, Belfort R Jr. Randomized clinical trial evaluating mETDRS versus normal or high-density micropulse photocoagulation for diabetic macular edema. Invest Ophthalmol Vis Sci. 2011 Jun 17;52(7):4314-23. doi: 10.1167/iovs.10-6828. PMID 21345996
- [Background] Venkatesh P, Ramanjulu R, Azad R, Vohra R, Garg S. Subthreshold micropulse diode laser and double frequency neodymium: YAG laser in treatment of diabetic macular edema: a prospective, randomized study using multifocal electroretinography. Photomed Laser Surg. 2011 Nov;29(11):727-33. doi: 10.1089/pho.2010.2830. Epub 2011 May 25. PMID 21612513
- [Background] Chen G, Tzekov R, Li W, Jiang F, Mao S, Tong Y. SUBTHRESHOLD MICROPULSE DIODE LASER VERSUS CONVENTIONAL LASER PHOTOCOAGULATION FOR DIABETIC MACULAR EDEMA: A Meta-Analysis of Randomized Controlled Trials. Retina. 2016 Nov;36(11):2059-2065. doi: 10.1097/IAE.0000000000001053. PMID 27096529
- [Background] Lupidi M, Coscas F, Cagini C, Coscas G. Optical Coherence Tomography Angiography in Macular Edema. Dev Ophthalmol. 2017;58:63-73. doi: 10.1159/000455269. Epub 2017 Mar 28. PMID 28351045
- [Background] Vujosevic S, Gatti V, Muraca A, Brambilla M, Villani E, Nucci P, Rossetti L, De Cilla' S. OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY CHANGES AFTER SUBTHRESHOLD MICROPULSE YELLOW LASER IN DIABETIC MACULAR EDEMA. Retina. 2020 Feb;40(2):312-321. doi: 10.1097/IAE.0000000000002383. PMID 31972802
- [Background] Cole ED, Novais EA, Louzada RN, Moult EM, Lee BK, Witkin AJ, Waheed NK, Duker JS, Baumal CR. Visualization of Changes in the Choriocapillaris, Choroidal Vessels, and Retinal Morphology After Focal Laser Photocoagulation Using OCT Angiography. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT356-61. doi: 10.1167/iovs.15-18473. PMID 27409493
- [Background] Tang FY, Ng DS, Lam A, Luk F, Wong R, Chan C, Mohamed S, Fong A, Lok J, Tso T, Lai F, Brelen M, Wong TY, Tham CC, Cheung CY. Determinants of Quantitative Optical Coherence Tomography Angiography Metrics in Patients with Diabetes. Sci Rep. 2017 May 31;7(1):2575. doi: 10.1038/s41598-017-02767-0. PMID 28566760
- [Background] Acon D, Wu L. Multimodal Imaging in Diabetic Macular Edema. Asia Pac J Ophthalmol (Phila). 2018 Jan-Feb;7(1):22-27. doi: 10.22608/APO.2017504. Epub 2017 Jan 29. PMID 29376234